CLINICAL TRIAL: NCT05105074
Title: Does the Use of Intrathecal Morphine Increase the Length of Hospital Stay in Fast Track Orthopedic Procedures?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Principal Investigator, Dr. Naveed Siddiqui, Associate Professor, Samuel Lunenfeld Research Institute, Mount Sinai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 18-0116-A
Record Dates: First submitted 2021-09-28; First posted 2021-11-03 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Arthropathy of Knee; Arthropathy of Hip
Keywords: Arthroplasty; Knee; Hip; Intrathecal Morphine; Urinary retention; Opioid
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal Morphine (Active Comparator): One group will receive intrathecal morphine 100 mcg in addition to the standard dose of bupivacaine and fentanyl 15 mcg for spinal anesthesia.
  Interventions: Drug: Intrathecal Morphine
- Placebo (Placebo Comparator): One group will receive normal saline 100 mcg in addition to the standard dose of bupivacaine and fentanyl 15 mcg for spinal anesthesia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intrathecal Morphine — Group 1 - Patients will receive intrathecal morphine 100 mcg in addition to the standard dose of bupivacaine and 15 mcg of fentanyl for spinal anesthesia.
  Arms: Intrathecal Morphine
Drug: Placebo — Group 2 - Patients will not receive intrathecal morphine. Patients will receive only bupivacaine and 15 mcg of fentanyl for spinal anesthesia.
  Arms: Placebo

SUMMARY:
This is a clinical trial of intrathecal morphine for patients Patient with primary as well as revision knee and hip arthroplasty under regional anesthesia. This study would include a total of 134 patients. It is the intention to randomize these patients postoperatively into 2 groups of patients:

Group 1 - Patients will receive intrathecal morphine 100 mcg in addition to the standard dose of bupivacaine and 15 mcg of fentanyl for spinal anesthesia.

Group 2 - Patients will not receive intrathecal morphine. Patients will receive only bupivacaine and 15 mcg of fentanyl for spinal anesthesia.

It is postulated that the use of intrathecal morphine may be associated with an increase length of stay in the hospital.

DETAILED DESCRIPTION:
Procedures:

Preoperative phase- The patients will receive the consent form together with the standard sheet in the pre-admission unit or remotely via telephone or email, usually one week before surgery, explaining intrathecal morphine and its benefits and drawbacks. These patients will receive an educational booklet regarding the "fast track protocol" which includes clear instruction related to their upcoming surgery. The material covers a wide range of topics such as instructions related to fasting for solids and liquids before coming for surgery, the expectation of pain relief and physiotherapy, types of anesthesia and expected length of hospital stay. Upon hospital admission, one hour before the procedure, patients will receive gabapentin 300mg, celecoxib 400mg (will be reduced to celecoxib 200mg in patients ≥ 65 years old) and acetaminophen 1000mg orally.

Intraoperative phase- Surgical procedures to be included in the study are elective primary as well as revision arthroplasty of knee and hip joints under spinal anesthesia with or without sedation. Patient will be randomized to one of two groups. One group will receive intrathecal morphine 100 mcg in addition to the standard dose of bupivacaine and fentanyl 15 mcg for spinal anesthesia and another group will not receive intrathecal morphine. Upon prosthesis implant, the surgeon will infiltrate periarticular 100 ml (40 ml bupivacaine 0.5% + 60 ml of normal saline) as per the orthopedic protocol. Sedation will be titrated to keeping modified Ramsay sedations score (RSS) between 3 and 5.

Postoperative phase- upon emergence from anesthesia patients will be taken to the recovery room. As per our hospital protocol, the patient will be catheterized if the bladder residual volume by ultrasound is 500ml or more. Post-operative pain score and opioid requirements and complications including urinary retention, vomiting and respiratory depression will be recorded. Overall duration of stay in the hospital will be noted. If any patient requires catheterization of bladder, the duration of catheter requirement and frequency of catheterization will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* Age 18 to 85 years
* BMI 18 to 40 kg/cm2
* Patient with primary as well as revision knee and hip arthroplasty under regional anesthesia only.
* Provision of written informed consent.

Exclusion Criteria:

* Language barrier or difficulty in communication: inability to read write or speak English
* Allergy to morphine
* Patients under increased risk for respiratory depression with intrathecal morphine (central apnea)
* Patients with pre-existing urinary problems
* Women of child bearing potential not on birth control
* Patients with chronic pain who are currently on pain medications
* Patients with cognitive impairment
* Patients who have alcohol and/or other substance dependency

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | From admission to the hospital until discharge, an average of 3 days
  Duration of stay in the hospital in hours

SECONDARY OUTCOMES:
Incidence of opioid related side effects | 48 Hours post operatively
  Nausea, Vomiting, Constipation, Difficulty passing urine, Difficulty concentrating, Dizziness, Drowsiness, Feeling confused, Fatigue, Itchiness, Dry mouth, Headache.
Time from Spinal Anesthesia to bladder catheterization | During the hospital admission, an average of 3 days
  Time from Spinal Anesthesia to bladder catheterization (Foley catheterization or In and Out catheterization ) in hours.
Pain scores measured at rest and movement twice a day | 48 Hours post operatively
  Based on Verbal Analogue Scale (VAS) scoring system (0-10), where score of 0 refers to no pain and a score of 10 refers to the worst pain imaginable
Overall feeling/ satisfaction about pain treatment | At the time of discharge from hospital, an average of 3 days
  Patient satisfaction from pain management during hospital stay, from score of 1(very dissatisfied) to score of 6 (Very satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Petros JG, Rimm EB, Robillard RJ. Factors influencing urinary tract retention after elective open cholecystectomy. Surg Gynecol Obstet. 1992 Jun;174(6):497-500. PMID 1350689
- [Background] Huang A, Ryu JJ, Dervin G. Cost savings of outpatient versus standard inpatient total knee arthroplasty. Can J Surg. 2017 Feb;60(1):57-62. doi: 10.1503/cjs.002516. PMID 28234591
- [Background] Murphy PM, Stack D, Kinirons B, Laffey JG. Optimizing the dose of intrathecal morphine in older patients undergoing hip arthroplasty. Anesth Analg. 2003 Dec;97(6):1709-1715. doi: 10.1213/01.ANE.0000089965.75585.0D. PMID 14633547
- [Background] David M, Arthur E, Dhuck R, Hemmings E, Dunlop D. High rates of postoperative urinary retention following primary total hip replacement performed under combined general and spinal anaesthesia with intrathecal opiate. J Orthop. 2015 Nov 18;12(Suppl 2):S157-60. doi: 10.1016/j.jor.2015.10.020. eCollection 2015 Dec. PMID 27047216
- [Background] Min BW, Kim Y, Cho HM, Park KS, Yoon PW, Nho JH, Kim SM, Lee KJ, Moon KH. Perioperative Pain Management in Total Hip Arthroplasty: Korean Hip Society Guidelines. Hip Pelvis. 2016 Mar;28(1):15-23. doi: 10.5371/hp.2016.28.1.15. Epub 2016 Mar 31. PMID 27536639
- [Background] McCartney CJ, McLeod GA. Local infiltration analgesia for total knee arthroplasty. Br J Anaesth. 2011 Oct;107(4):487-9. doi: 10.1093/bja/aer255. No abstract available. PMID 21903643
- [Background] Jia XF, Ji Y, Huang GP, Zhou Y, Long M. Comparison of intrathecal and local infiltration analgesia by morphine for pain management in total knee and hip arthroplasty: A meta-analysis of randomized controlled trial. Int J Surg. 2017 Apr;40:97-108. doi: 10.1016/j.ijsu.2017.02.060. Epub 2017 Feb 24. PMID 28254422